CLINICAL TRIAL: NCT07241065
Title: An Open-label, Fixed-sequence Study to Assess the Effect of Capivasertib on the Pharmacokinetics of Oral Dextromethorphan (CYP2D6 Substrate) in Healthy Participants.
Brief Title: A Study to Investigate the Effect of Capivasertib on the Pharmacokinetics of Oral Dextromethorphan (CYP2D6 Substrate) in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: D3615C00005
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Serine/protein kinase AKT; Anti-cancer agent; Pharmacokinetics; Protein kinase
MeSH Terms: interventions — Dextromethorphan; capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dextromethorphan/ Dextromethorphan + Capivasertib (Experimental): Participants will receive a single dose of dextromethorphan in Period 1. After a minimum washout period of 4 days from the first dose of dextromethorphan, participants will receive the first dose of capivasertib, followed by a second dose of capivasertib after 12 hours, administered concomitantly with a single dose of dextromethorphan in Period 2.
  Interventions: Drug: Dextromethorphan; Drug: Capivasertib

INTERVENTIONS:
Drug: Dextromethorphan — Dextromethorphan will be administered orally once in Period 1 and once in Period 2
Drug: Capivasertib — Capivasertib will be administered orally twice in Period 2

SUMMARY:
The purpose of this study is to assess the effect of capivasertib on the pharmacokinetics of oral dextromethorphan in healthy participants.

DETAILED DESCRIPTION:
This is an open-label, fixed sequence study conducted at a single study centre.

The study will comprise of:

* A Screening Period (from Day -28 to Day -2)
* In-house treatment period (from Day -1 to Day 8) Period 1 (from Day -1 to Day 3): Participants will receive single oral doses of dextromethorphan during this period.

Period 2 (from Day 4 to Day 8): Participants will receive 2 doses of capivasertib and a single dose of dextromethorphan during this period.

• Follow-up Visit within 7 to 10 days after the last administration of the Investigative Medical Products (from Day 13 to Day 16).

ELIGIBILITY:
Main Inclusion Criteria:

* Have a Body Mass Index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg.
* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of non-childbearing potential must be confirmed at the screening visit (postmenopausal or documentation of irreversible surgical sterilisation).
* Male participants must have documentation of vasectomy done 6 months prior to screening visit. Participants must be willing to use one barrier method of contraception (condom) during sexual intercourse with a female partner of childbearing potential from the time of first study intervention administration until 16 weeks after the last dose of capivasertib.

Main Exclusion Criteria:

* History of any clinically important disease or disorder
* History or presence of gastrointestinal, hepatic or renal disease.
* Any clinically important illness, medical/surgical procedure (excluding placement of vascular access), or significant traumatic injury within 4 weeks of the first administration of study intervention or an anticipated need for major surgery during the study.
* Any clinically significant skin abnormalities that are chronic or currently active.
* Abnormal hepato-renal and bone marrow organ function laboratory values.
* Any clinically important abnormalities in clinical chemistry, haematology, or urinalysis.
* Any clinically significant abnormalities in glucose metabolism.
* Any positive result on screening for serum HBsAg OR anti-HBc antibody, indicative of active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Current smokers or those who have smoked or used other nicotine/nicotine-containing products within the previous 3 months prior to Screening Visit.
* Known or suspected history of alcohol or drug abuse or excessive intake of alcohol.
* Use of drugs with enzyme inducing properties 3 weeks prior to the first administration of study intervention.
* Use of strong inhibitors of Cytochrome P450 3A4 (CYP3A4) or strong/moderate inducers of CYP3A4 within 2 weeks prior to first dose of capivasertib.
* Concurrent use of herbal or natural products intended as treatment or prophylaxis that may interact with capivasertib.
* Participants who have previously received capivasertib.
* Any clinically significant abnormal findings in vital signs and 12-lead electrocardiogram (ECG).
* History of severe allergy/hypersensitivity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-12-03 (Estimated); Study Completion 2027-12-03 (Estimated)

PRIMARY OUTCOMES:
Area under concentration time curve from time 0 to infinity (AUCinf) of dextromethorphan | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (AUCinf) of dextromethorphan when administered orally alone and following oral dosing of capivasertib
Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) of dextromethorphan | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (AUClast) of dextromethorphan when administered orally alone and following oral dosing of capivasertib
Maximum observed drug concentration (Cmax) of dextromethorphan | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (Cmax) of dextromethorphan when administered orally alone and following oral dosing of capivasertib

SECONDARY OUTCOMES:
Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) of capivasertib | Period 2: Day 5 to Day 8
  To evaluate the PK (AUClast) of capivasertib following oral dosing
Time to reach maximum observed concentration (tmax) of capivasertib | Period 2: Day 5 to Day 8
  To evaluate the PK (tmax) of capivasertib following oral dosing
Maximum observed drug concentration (Cmax) of capivasertib | Period 2: Day 5 to Day 8
  To evaluate the PK (Cmax) of capivasertib following oral dosing
Ratio of AUCinf following co-administration to AUCinf following dosing alone (R AUCinf) of dextromethorphan | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (R AUCinf) of dextromethorphan following oral dosing
Ratio of AUClast following co-administration to AUClast following dosing alone (R AUClast) of dextromethorphan | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (R AUClast) of dextromethorphan following oral dosing
Ratio of Cmax following co-administration to Cmax following dosing alone (R Cmax) of dextromethorphan | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (R Cmax) of dextromethorphan following oral dosing
Terminal elimination half-life (t1/2λz) of dextromethorphan | Period 1: Day 1 to Day 3
  To evaluate the PK (t1/2λz) of dextromethorphan following oral dosing
Terminal rate constant (λz) of dextromethorphan | Period 1: Day 1 to Day 3
  To evaluate the PK (λz) of dextromethorphan following oral dosing
Time to reach maximum observed concentration (tmax) of dextromethorphan | Period 1: Day 1 to Day 3
  To evaluate the PK (tmax) of dextromethorphan following oral dosing
Area under concentration time curve from time 0 to infinity (AUCinf) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3
  To evaluate the PK (AUCinf) of dextromethorphan following oral dosing
Area under concentration curve from time 0 to the last quantifiable concentration (AUClast) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3
  To evaluate the PK (AUClast) of dextromethorphan following oral dosing
Maximum observed drug concentration (Cmax) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3
  To evaluate the PK (Cmax) of dextromethorphan following oral dosing
Ratio of AUClast following co-administration to AUClast following dosing alone (R AUClast) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3, Period 2: Day 6 to Day 8
  To evaluate the PK (R AUClast) of dextromethorphan following oral dosing
Terminal elimination half-life (t1/2λz) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3
  To evaluate the PK (t1/2λz) of dextromethorphan following oral dosing
Terminal rate constant (λz) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3
  To evaluate the PK (λz) of dextromethorphan following oral dosing
Time to reach maximum observed concentration (tmax) of metabolite (dextrorphan) | Period 1: Day 1 to Day 3
  To evaluate the PK (tmax) of dextromethorphan following oral dosing
Number of participants with adverse events (AEs) and serious AEs | Up to Day 16
  To examine the safety and tolerability of capivasertib when administered with dextromethorphan
Percentage change from baseline in bilirubin levels | Period 1: Day 1 to Day 2, Period 2: Day 4 to Day 7
  To evaluate the effect of capivasertib dosing on total, conjugated, and unconjugated bilirubin levels

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/